CLINICAL TRIAL: NCT01993095
Title: Improving Functional Performance in Persons With MS Via Physical Activity DVD Intervention
Brief Title: FlexToBa for People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Edward McAuley, Professor, Kinesiology and Community Health, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IL-0009
Record Dates: First submitted 2013-10-18; First posted 2013-11-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Quality of Life; Functional Fitness
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: FlexToBa physical activity DVD (Experimental): Participants in this arm will receive a physical activity program delivered by DVD that focuses on exercises targeting flexibility, toning and balance. These exercises will be progressive in nature throughout the six months and will also focus on modifications for all ability levels. Participants will be provided with three DVDs including: an Introduction to physical activity, Sessions 1-3, and Sessions 4-6, which they will be asked to watch and participate in over the course of six months.
  Interventions: Behavioral: Home-based, DVD-delivered physical activity
- Usual care-Wait list (Active Comparator): Participants in this arm will receive a DVD that focuses on healthy aging topics but does not include physical activity. They will receive the FlexToBa DVD after the completion of the 6-month follow-up testing.
  Interventions: Behavioral: Behavioral: Usual care/Wait list

INTERVENTIONS:
Behavioral: Home-based, DVD-delivered physical activity — Subjects will be participating in a home-based physical activity program that focuses on flexibility, toning and balance. Exercises will be progressive over the six-months and will highlight modifications for varying levels. This program will be delivered on 3 DVDs. Participants will be asked to exercise with the DVD at least three times per week.
  Arms: Experimental: FlexToBa physical activity DVD
Behavioral: Behavioral: Usual care/Wait list — Participants in this arm will receive a DVD that focuses on healthy aging topics but does not include physical activity. They will receive the FlexToBa DVD after the completion of the 6-month follow-up testing.
  Arms: Usual care-Wait list

SUMMARY:
The purpose of this study is to test the effectiveness of a DVD-delivered, home-based six-month physical activity intervention for people with Multiple Sclerosis.

DETAILED DESCRIPTION:
Persons with MS are less likely to be active than their healthy counterparts, a statistic that is compounded by the symptom manifestations of MS. However, there is increasing evidence to support the importance of physical activity in MS. Unfortunately, structured, safe, and efficacious physical activity programs that are often conducted in medical or university settings are often not accessible to many older adults with or without MS. We propose to conduct a randomized controlled pilot trial testing the efficacy of a DVD-delivered physical activity intervention which targets factors that have the potential to reduce disability in older adults with MS. This DVD-based intervention has been previously approved by the IRB at the University of Illinois for a similar study with low-active, community-dwelling older adults (IRB Protocol Number: 09765). This novel intervention provides systematic, programmatic activities with alternative versions of each exercise that allow individuals of all capabilities to complete the program successfully. It focuses on improving flexibility, strength, and balance and has been demonstrated to be feasible, well-accepted, and efficacious in a large sample of older adults without MS. Importantly, intervention resulted in clinically significant improvements in the Short Physical Performance Battery, reliable determinant of disability, institutionalization, morbidity, and mortality. If such an intervention was equally successful in older persons with MS, this could have considerable public health impact.

ELIGIBILITY:
Inclusion Criteria:

* being non-active, defined as reporting not engaging in regular activity (30 minutes accumulated per day) on more than two days of the week in the prior six months;
* aged 50 years and older;
* fluent in English;
* relapse-free in the last 30 days;
* ambulatory with minimal assistance(i.e., walk independently or with a single-point assistive walking device such as a cane);
* the provision of medical clearance for participation in a physical activity program by participants' physicians, along with a physician-confirmed diagnosis of MS (communication with physicians will be facilitated by research staff).

Exclusion Criteria:

* self-reported physical activity on a regular basis within the last six months (2 times or more per week);
* younger than 50 years of age;
* relapse in the last 30 days;
* no regular access to a television;
* no physician-confirmed diagnosis of multiple sclerosis;
* unable to successfully score above 21 (out of 39)on the Telephone Interview of Cognitive Status questionnaire (TICS-M).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to six-months in assessments of functional fitness of sedentary adults who have Multiple Sclerosis | Baseline and six months
  The measurements will include:
  Short physical performance battery -- measures walking speed, ability to rise from a chair, and standing balance
Change from baseline to six-months in assessments of functional fitness of sedentary adults who have MS | Baseline and six-months
  Measurements will include:
  Timed 20-foot walk test -- walk 25 feet as quickly as possible;
Change in assessments of functional fitness assessments in sedentary adults with MS | Baseline and six-months
  Measurements will include:
  6-minute walk test -- walk as much as possible (in terms of distance) for 6 minutes;
Change from baseline to six-months in assessments of functional fitness of sedentary adults with MS | Baseline and six-months
  Measurements will include:
  Grip strength -- using a dynamometer, participants will demonstrate isometric grip strength;
Change from baseline to six-months in assessments of functional fitness of sedentary adults who have MS | Baseline and six-months
  Measurements will include:
  Flexibility -- sit and reach (lower body flexibility) and back scratch test (upper body flexibility)
Change from baseline to six-months in assessments of functional fitness of sedentary adults with MS | Baseline and six-months
  Measurements will include:
  Upper body strength -- bicep curls consisting of lifting a light hand-weight as many times as possible in 30-seconds;
Change from baseline to six-months in assessments of functional fitness of sedentary adults who have MS | Baseline and six-months
  Measurements will include:
  Balance -- a timed (up to 30-seconds) unassisted one-leg stand test with eyes open on each leg.
Change from baseline to six-months in assessments of reported quality of life in people with MS | Baseline and six months
  The Leeds Multiple Sclerosis Quality of Life Scale will be used as a disease specific quality of life measure for people with MS.
Change from baseline to six-months in assessments of reported quality of life in people with MS | Baseline and six-months
  The Satisfaction with Life Scale will be used to assess global life satisfaction and is sensitive enough to detect changes in participants' perceptions over the course of a clinical intervention.

SECONDARY OUTCOMES:
Change from baseline to six-months in assessments of cognitive performance in sedentary adults with MS | Baseline and six months
  The Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) battery, which will be administered to assess cognitive performance.
Change from baseline to six-months in assessments of reported barriers self-efficacy in people with MS | Baseline and six months
  Participants' situation-specific self-confidence for physical activity will be assessed using The Barriers Self-Efficacy Scale, which taps subjects' perceived capabilities to exercise three times per week for 40 minutes over the next two months in the face of commonly identified barriers to participation.
Changes in physical activity relating to specified exercise program in sedentary adults with MS | Baseline and six months
  Adherence to exercise program as documented by daily exercise logs.
Objective changes in physical activity in sedentary adults with MS | Baseline and six months
  Objective assessment of physical activity via accelerometry over seven days time.
Self-reported changes in physical activity in sedentary adults with MS | Baseline and six months
  Subjective assessment of physical activity via the Godin Leisure Time Exercise Questionnaire, which assesses frequency of involvement in strenuous, moderate and light activities.
Change from baseline to six-months in assessments of reported gait self-efficacy in sedentary adults with MS | Baseline and six-months
  Participants' situation-specific self-confidence for physical activity will be assessed using The Gait Self-Efficacy Scale, which will assess participants' beliefs in their capabilities to negotiate stairs and objects in their path.
Change from baseline to six-months in assessments of reported exercise self-efficacy in sedentary people with MS | Baseline and six-months
  The Exercise Self-Efficacy Scale will assess participants' beliefs in their ability to continue exercising on a three time per week basis at moderate intensities for 40+ minutes per session in the future.
Change from baseline to six-months in assessments of reported self-efficacy of walking in sedentary people with MS | Baseline and six-months
  Walking Self-Efficacy Scale for Duration will assess participants' beliefs in their physical capability to successfully complete incremental 5-minute intervals (up to 40 minutes)of walking at a moderately fast pace.

CONTACTS AND LOCATIONS:
Overall Officials: Edward McAuley, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wojcicki TR, Roberts SA, Learmonth YC, Hubbard EA, Kinnett-Hopkins D, Motl RW, McAuley E. Improving physical functional and quality of life in older adults with multiple sclerosis via a DVD-delivered exercise intervention: a study protocol. BMJ Open. 2014 Dec 1;4(12):e006250. doi: 10.1136/bmjopen-2014-006250. PMID 25448627
- See also: Exercise Psychology Lab at University of Illinois at Urbana-Champaign — http://www.epl.illinois.edu